CLINICAL TRIAL: NCT01247064
Title: Nebulized Hypertonic Saline for Acute Bronchiolitis in the Emergency Department
Brief Title: Hypertonic Saline for Acute Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 10-007460
Record Dates: First submitted 2010-11-15; First posted 2010-11-24 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Bronchiolitis, Viral; Saline Solution, Hypertonic
Keywords: Bronchiolitis; Hypertonic Saline
MeSH Terms: conditions — Bronchiolitis, Viral; Bronchiolitis | interventions — Sodium Chloride; Saline Solution, Hypertonic; Inhalation; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulized 3% Saline (Experimental)
  Interventions: Drug: Nebulized 3% saline
- Nebulized 0.9% Normal Saline (Placebo Comparator)
  Interventions: Drug: Nebulized 0.9% Normal Saline

INTERVENTIONS:
Drug: Nebulized 3% saline — 4 mL of nebulized 3% saline once
  Other Names: 3% Hypertonic Saline Solution for Inhalation
  Arms: Nebulized 3% Saline
Drug: Nebulized 0.9% Normal Saline — 4 mL of 0.9% nebulized normal saline once
  Other Names: 0.9% Saline Solution for Inhalation
  Arms: Nebulized 0.9% Normal Saline

SUMMARY:
The purpose of this study is to determine whether nebulized 3% hypertonic saline (HS) improves respiratory distress in children 2-23 months presenting to the emergency department (ED) with acute bronchiolitis with persistent respiratory distress after initial therapy with a trial of nebulized albuterol.

DETAILED DESCRIPTION:
Acute bronchiolitis is the most frequent cause of infant hospitalization in the United States. Bronchiolitis typically refers to a viral lower respiratory tract infection during the first two years of life manifesting as a constellation of clinical symptoms including wheezing, cough and respiratory distress. In addition to a tremendous disease burden, bronchiolitis admissions in the United States cost more than $500 million each year.

The primary pathophysiologic processes in bronchiolitis include airway wall and peribronchial inflammation, increased mucous production, sloughing of necrotic epithelial cells, and impaired airway clearance. These processes result in airway obstruction, gas trapping, atelectasis and impaired gas exchange. Standard therapies for bronchiolitis remain supportive, including maintaining hydration and nutrition, ensuring adequate oxygenation, and physical suctioning of the nasal airways to clear secretions. Therapies such as the bronchodilator albuterol, although commonly used in standard practice, have not been proven to impact progression of disease or improve long-term outcomes of bronchiolitis.

Nebulized hypertonic saline (HS) has been shown to increase mucociliary clearance in the airways of individuals with healthy lungs. In addition nebulized HS increases airway clearance for disease processes including asthma, cystic fibrosis and bronchiectasis. A recent Cochrane review examined 4 small studies that suggest that nebulized 3% HS may reduce length of hospital stay and improve clinical severity scores in infants with acute viral bronchiolitis. None of these studies have explored the use of nebulized HS in the emergency department (ED). A recent study examined the use of a single nebulized treatment of epinephrine mixed in 3% HS in 46 infants less than 12 months presenting to the ED with bronchiolitis. This study did not find a difference between epinephrine diluted in normal saline compared to epinephrine diluted in 3% HS. Despite no effect on clinical score, the investigators did note a trend toward decreased rates of hospitalization. Furthermore, since this was the first ED study and the first negative study, the authors concluded that further investigation is necessary to determine if HS has a role in the management of acute bronchiolitis.

The purpose of the current study is to determine whether nebulized 3% HS improves respiratory distress in children 2-23 months presenting to the ED with acute bronchiolitis with persistent respiratory distress after initial therapy with a trial of nebulized albuterol.

Given the tremendous clinical and financial burden of bronchiolitis, any effective therapy, particularly one that is inexpensive, has the potential to result in significant health care savings. If nebulized 3% HS improved clinical scores in the ED, this may provide an inexpensive, safe and effective therapy for children with bronchiolitis in the acute care setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 weeks through 23 months
* First episode of wheezing associated with respiratory distress and upper respiratory tract infection.
* Respiratory Distress Assessment Instrument (RDAI) rating of ≥4 and ≤15 after initial albuterol nebulization per standard care
* Pediatric Emergency Medicine (PEM) physician does not plan additional bronchodilator therapy within the hour after initial assessment.
* Parental/guardian permission (informed consent)

Exclusion Criteria:

* Subjects with prior history of wheezing or asthma or who have received bronchodilator therapy prior to the current illness
* Chronic lung or heart disease
* Critically ill infants requiring immediate airway stabilization
* Non-English speaking parent/guardian
* Inability to take nebulized medications

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zorc, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Todd Florin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Grewal S, Ali S, McConnell DW, Vandermeer B, Klassen TP. A randomized trial of nebulized 3% hypertonic saline with epinephrine in the treatment of acute bronchiolitis in the emergency department. Arch Pediatr Adolesc Med. 2009 Nov;163(11):1007-12. doi: 10.1001/archpediatrics.2009.196. PMID 19884591
- [Background] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulized hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006458. doi: 10.1002/14651858.CD006458.pub2. PMID 18843717
- [Background] Kuzik BA, Al-Qadhi SA, Kent S, Flavin MP, Hopman W, Hotte S, Gander S. Nebulized hypertonic saline in the treatment of viral bronchiolitis in infants. J Pediatr. 2007 Sep;151(3):266-70, 270.e1. doi: 10.1016/j.jpeds.2007.04.010. Epub 2007 Jun 29. PMID 17719935
- [Background] Tal G, Cesar K, Oron A, Houri S, Ballin A, Mandelberg A. Hypertonic saline/epinephrine treatment in hospitalized infants with viral bronchiolitis reduces hospitalization stay: 2 years experience. Isr Med Assoc J. 2006 Mar;8(3):169-73. PMID 16599051
- [Background] Mandelberg A, Tal G, Witzling M, Someck E, Houri S, Balin A, Priel IE. Nebulized 3% hypertonic saline solution treatment in hospitalized infants with viral bronchiolitis. Chest. 2003 Feb;123(2):481-7. doi: 10.1378/chest.123.2.481. PMID 12576370
- [Background] Sarrell EM, Tal G, Witzling M, Someck E, Houri S, Cohen HA, Mandelberg A. Nebulized 3% hypertonic saline solution treatment in ambulatory children with viral bronchiolitis decreases symptoms. Chest. 2002 Dec;122(6):2015-20. doi: 10.1378/chest.122.6.2015. PMID 12475841
- [Derived] Florin TA, Shaw KN, Kittick M, Yakscoe S, Zorc JJ. Nebulized hypertonic saline for bronchiolitis in the emergency department: a randomized clinical trial. JAMA Pediatr. 2014 Jul;168(7):664-70. doi: 10.1001/jamapediatrics.2013.5306. PMID 24862342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.2 (5.1) | 6.1 (3.6) | 6.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 24 | 23 | 47
  White | 3 | 3 | 6
  Hispanic | 1 | 5 | 6
  Asian | 2 | 0 | 2
  Missing | 1 | 0 | 1
Eczema History [Number; unit: participants]
  Yes | 8 | 7 | 15
  No | 21 | 23 | 44
  Unknown | 2 | 1 | 3
Family History of Atopy [Number; unit: participants]
  No | 7 | 6 | 13
  Yes | 22 | 24 | 46
  Unknown | 2 | 1 | 3
Days of Symptoms [Mean (Standard Deviation); unit: days] | 3.4 (3.7) | 3.4 (2.4) | 3.4 (3.1)
Smokers in Household [Number; unit: participants]
  No | 14 | 17 | 31
  Yes | 17 | 13 | 30
  Unknown | 0 | 1 | 1
ICU History [Number; unit: participants]
  No | 23 | 27 | 50
  Yes | 6 | 4 | 10
  Unknown | 2 | 0 | 2
Respiratory Distress Assessment Instrument Score [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0 to 17. Higher values indicate worse respiratory distress.
  units on a scale | 7.8 (2.6) | 7.4 (2.5) | 7.6 (2.5)
Respiratory Rate [Mean (Standard Deviation); unit: breaths per minute] | 49.6 (12.4) | 52.4 (12.4) | 50.9 (12.3)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 153.4 (18.4) | 159.3 (21.9) | 156.5 (20)
Oxygen Saturation [Mean (Standard Deviation); unit: percent] | 95.4 (3.8) | 96.3 (3.7) | 95.9 (3.7)
Physician Clinical Impression [Number; unit: participants]
  Mild | 9 | 11 | 20
  Moderate | 21 | 20 | 41
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Assessment Change Score (RACS)
Description: The Respiratory Assessment Change Score (RACS) assesses change in respiratory status using the change in the Respiratory Distress Assessment Instrument (RDAI) and a standardized change in respiratory rate, with points being assigned by change increments of 10%. Thus, a change in respiratory rate of ≤5% from baseline counted as a change of 0 units, decrease/increase of 6% to 15% counted as improvement/deterioration of 1 unit, etc. The overall RACS is the arithmetic sum of the RDAI change and the standardized respiratory rate change between assessments with a decrease in RACS signifying improvement.
Time Frame: Baseline and 1 hour
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Number analyzed (Participants) | 31 | 31
units on a scale | -1.5 [-3.1 to 0.2] | -4 [-5.3 to -2.7]
Statistical Analysis 1: Comparison: Nebulized 3% Saline vs Nebulized 0.9% Normal Saline; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

2. Secondary Outcome: Rate of Hospitalization
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Number analyzed (Participants) | 31 | 31
percentage of participants | 71 | 64.5
Statistical Analysis 1: Comparison: Nebulized 3% Saline vs Nebulized 0.9% Normal Saline; Test type: Superiority or Other; p = 0.86, Chi-squared

3. Secondary Outcome: Respiratory Rate Change
Time Frame: Baseline and 1 hour
Measure: Mean (95% Confidence Interval); unit: breaths per minute
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Number analyzed (Participants) | 31 | 31
breaths per minute | -1.8 [-6.5 to 2.8] | -9.8 [-14.6 to -4.9]
Statistical Analysis 1: Comparison: Nebulized 3% Saline vs Nebulized 0.9% Normal Saline; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

4. Secondary Outcome: Oxygen Saturation Change
Time Frame: Baseline and 1 hour
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Number analyzed (Participants) | 31 | 31
percent | 1.1 [-0.4 to 2.6] | 0.1 [-1.6 to 1.8]
Statistical Analysis 1: Comparison: Nebulized 3% Saline vs Nebulized 0.9% Normal Saline; Test type: Superiority or Other; p = 0.36, t-test, 2 sided

5. Secondary Outcome: Parental Perception of Improvement of Breathing After Study Medication
Time Frame: 1 hour
Measure: Number; unit: percentage of participants
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Number analyzed (Participants) | 31 | 31
percentage of participants | 50 | 54.8
Statistical Analysis 1: Comparison: Nebulized 3% Saline vs Nebulized 0.9% Normal Saline; Test type: Superiority or Other; p = 0.62, Chi-squared

ADVERSE EVENTS:
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes